CLINICAL TRIAL: NCT06643637
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Multiple Doses of MLS101 (Psilocybin) in Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Multiple Doses of MLS101 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MycoMedica Life Sciences PBC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-MLS101-102
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled multiple dose study to assess the safety, tolerability, and pharmacokinetics of MLS101 in healthy participants.
  Multiple Dose (MD): 16 participants will be enrolled in two dose cohorts and will be randomized to receive multiple doses of MLS101 or placebo. An additional cohort (8 participants) may enrolled to explore more doses.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MLS101 (Active Comparator): MLS101 capsule(s) administered orally as a once a day dose
  Interventions: Drug: Psilocybin
- Placebo (Placebo Comparator): Active treatment matching capsules will be administered orally as a once a day dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin — Capsule containing active ingredient, psilocybin
  Other Names: MLS101
  Arms: MLS101
Drug: Placebo — Capsule with no active ingredients
  Arms: Placebo

SUMMARY:
MLS101 is being developed as a low dose psilocybin, that can be administered to treat neurological and psychiatric conditions.

The purpose of this clinical trial is to assess how safe and tolerated MLS101 is; to see how MLS101 is distributed and cleared by the body (pharmacokinetics); and to assess the psychedelic effects of MLS101 in healthy, adult participants.

DETAILED DESCRIPTION:
In recent years, high-dose psilocybin has gained attention for it potential therapeutic benefit in many psychiatric conditions, however existing clinical data for low psilocybin doses are limited.

Microdoses are generally considered to be those absent of profound sensory and cognitive effects that would interfere with normal everyday functioning, but only a small number of prospective studies have evaluated microdoses and/or low doses in a controlled manner.

As a foundational study of the therapeutic use of psilocybin microdoses, this study will assess the safety, tolerability, pharmacokinetics and sensorial effects using a prospective, controlled, multiple dose regimen in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 to 65 years old (inclusive) at the time of signing the informed consent form. Standard contraception measures are required for this clinical trial.
2. Healthy, in the opinion of the Investigator, based on prior (history of) or current (ongoing) medical and psychiatric screening assessments.
3. Participants with no clinically significant findings on physical examination, laboratory tests, and cardiac assessment.
4. Body mass index (BMI) within the range 18-32 kg/m2, inclusive.
5. Normal blood pressure.
6. Capable of giving signed informed consent which includes the requirements and restrictions as per the approved study protocol.

Exclusion Criteria:

1. Prior known exposure to psilocybin within the past 5 years.
2. Prior (history of) or current (ongoing) diagnosis, or first-degree relatives with clinically significant medical or psychiatric condition or disease.
3. History of or presence of cardiovascular disease.
4. Abnormal and clinically significant ECG.
5. History or presence of a neurodegenerative disorder such Alzheimer's disease or Parkinson's disease.
6. Use of medications that have CNS effects or affect performance.
7. Use of medications with serotonergic activity.
8. History or presence of hypersensitivity or idiosyncratic reaction to psilocybin or related compounds.
9. History of substance or alcohol abuse disorder in the last 1 year.
10. Participant who, for any reason, is deemed by the Investigator to be inappropriate for this study; or has any condition which would confound or interfere with the evaluation of the safety, tolerability, or PK of the investigational drug; or is unable to comply with the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and seriousness of treatment-emergent adverse events (TEAEs) | Screening (Day -28) to end of study visit (Cohort 1: Day 15; Cohort 2: Day 23)
  Physical examinations, safety laboratory tests, ECGs
Occurrence of clinically significant changes in physical examination, vital signs, ECGs, clinical laboratory tests, the Columbia-Suicide Severity Rating Scale (C-SSRS). | Screening (Day -28) to end of study visit (Cohort 1: Day 15; Cohort 2: Day 23)
  The Columbia Suicide Severity Rating Scale (C-SSRS) is a short questionnaire. If there is a positive result for suicidality on the C-SSRS after Screening (defined by a participant answering "yes" to questions 4 or 5 on the suicidal ideation portion of the C-SSRS), the participant will be evaluated by an Investigator or medically qualified Sub-investigator for continuation in the study. Participants with suicidal ideation or behaviour (a "yes" answer at any time during treatment to any one of the ten suicidal ideation and behaviour questions (Categories 1-10) on the C-SSRS) at any time during the study will be withdrawn from the study. If a participant becomes suicidal during the study, an Investigator or medically qualified Sub-investigator should provide the appropriate treatment to the participant.

SECONDARY OUTCOMES:
Pharmacokinetics of MLS101: maximum observed serum concentration (Cmax) | Day 1 to Day 8 pre-dose, Day 1 to Day 9 post-dose (Cohort 1); Day 1 to Day 16 pre-dose, Day 1 to Day 17 post-dose (Cohort 2)
  Blood sample collections
Pharmacokinetics of MLS101: area under the plasma concentration-time curve (AUC) | Day 1 to Day 8 pre-dose, Day 1 to Day 9 post-dose (Cohort 1); Day 1 to Day 16 pre-dose, Day 1 to Day 17 post-dose (Cohort 2)
  Blood sample collections
Pharmacokinetics of MLS101: time corresponding to the occurrence of Cmax (Tmax) | Day 1 to Day 8 pre-dose, Day 1 to Day 9 post-dose (Cohort 1); Day 1 to Day 16 pre-dose, Day 1 to Day 17 post-dose (Cohort 2)
  Blood sample collections
Pharmacokinetics of MLS101: apparent terminal elimination half-life (t½) | Day 1 to Day 8 pre-dose, Day 1 to Day 9 post-dose (Cohort 1); Day 1 to Day 16 pre-dose, Day 1 to Day 17 post-dose (Cohort 2)
  Blood sample collections
Pharmacokinetics of MLS101: apparent total systemic clearance after oral administration (CL/F) | Day 1 to Day 8 pre-dose, Day 1 to Day 9 post-dose (Cohort 1); Day 1 to Day 16 pre-dose, Day 1 to Day 17 post-dose (Cohort 2)
  Blood sample collections
Pharmacokinetics of MLS101: apparent volume of distribution during the terminal phase (Vz/F) | Day 1 to Day 8 pre-dose, Day 1 to Day 9 post-dose (Cohort 1); Day 1 to Day 16 pre-dose, Day 1 to Day 17 post-dose (Cohort 2)
  Blood sample collections
Sensorial effects of MLS101 | Day 1 to Day 8 pre- and post-dose (Cohort 1); Day 1 to Day 16 pre- and post-dose (Cohort 2)
  Using validated questionnaires, the nominal sensorial threshold dose of MLS101 will be identified. The nominal sensorial threshold dose is defined as the highest dose studied that is absent of clinically significant sensorial effects, and which would not interfere with the participant's ability to carry on with routine activities of daily living. Higher scores indicate presence of sensorial effects.
Cognitive function: Digit Symbol Substitution Test (DSST) | Pre-dose (Day -1), Day 1, Day 4 and Day 8 (Cohort 1); Pre-dose (Day -1), Day 1, Day 4 and Day 16 (Cohort 2)
  The test taker's score is the number of correct symbol-to-number matches they complete within the allotted time.
Cognitive Function: Stroop Color and Word Test (SCWT) | Pre-dose (Day -1), Day 1, Day 4 and Day 8 (Cohort 1); Pre-dose (Day -1), Day 1, Day 4 and Day 16 (Cohort 2)
  Participants read tables of words and colors as quickly as possible.
Cognitive function: Trail Making Test A (TMT-A) | Pre-dose (Day -1), Day 1, Day 4 and Day 8 (Cohort 1); Pre-dose (Day -1), Day 1, Day 4 and Day 16 (Cohort 2)
  The participant draws lines to connect circled numbers in an ascending pattern (i.e., in numerical sequence 1-2-3, etc.) as rapidly as possible. The score is the time it takes the participant to complete the task in seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia